CLINICAL TRIAL: NCT05789199
Title: Retrospective Analysis of Real-World Use of Cefiderocol in the Management of Gram-Negative Infections as Part of the Early Access Program (PERSEUS Study)
Brief Title: Use of Cefiderocol in the Management of Gram-Negative Infections
Acronym: PERSEUS
Status: Completed | Type: Observational
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Other Study IDs: 2020-266-4
Record Dates: First submitted 2023-02-16; First posted 2023-03-29 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Gram-Negative Infection
Keywords: Cefiderocol; Early Access Program; Spain
MeSH Terms: interventions — Cefiderocol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Microbiological samples representative of the infection, when available, will be sent by investigating sites to a third party for characterization and analysis. The results of this microbiological characterization will be inputted into the database linked to the participant episode via the electronic study case record form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cefiderocol Treated: Participants who have been treated with at least 72 hours of cefiderocol through the EAP in Spain.
  Interventions: Drug: Cefiderocol

INTERVENTIONS:
Drug: Cefiderocol — Cefiderocol is a novel siderophore cephalosporin developed for the treatment of infections caused by Gram-negative bacteria (GNB), including those resistant to carbapenems.

SUMMARY:
The aim of this study is to describe the use of cefiderocol in the management of Gram-negative infections (GNIs) in participants treated through the Early Access Program (EAP) in Spain.

DETAILED DESCRIPTION:
This is a multicenter, retrospective, chart review of existing medical records in participants who received cefiderocol for a GNI as part of the Shionogi EAP. Access to cefiderocol was granted as Medication not approved in Spain subject to RD 1015/2009, which dictates that each case is approved on an individual basis by the Spanish Agency of Medicines. This study will be conducted at Spanish sites where cefiderocol was supplied via the EAP, beginning in 2018.

ELIGIBILITY:
Inclusion Criteria:

* Have received first course of cefiderocol.
* Have received treatment for at least 72 hours (complete) with cefiderocol as a part of clinical compassionate management, requested in the EAP.

Exclusion Criteria:

* Enrolled in any clinical trial of an investigational product.
* Documented Acinetobacter spp infection.
* Incomplete medical records for the following essential data elements:
* Cefiderocol usage (dose, duration, frequency)
* Data to be able to determine clinical success (primary objective)
* Co-infection with a GNB resistant to cefiderocol in 28 days of the initial dose of cefiderocol.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants treated with cefiderocol for GNIs through the EAP in Spain.
Sampling Method: Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2022-07-31 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Rate Of Clinical Success | From Day 1 (cefiderocol initiation) through Day 28
  The rate of clinical success will be reported as the percent clinical success of participants treated with cefiderocol for participants who receive at least 72 hours of cefiderocol through the EAP for the treatment of Gram-negative, carbapenem-resistant infections (except for Acinetobacter spp).

SECONDARY OUTCOMES:
Number of Participants Experiencing Resolution of Infection or Clinical Cure After Treatment With Cefiderocol | Day 1 (cefiderocol initiation), every 7 days up to Day 28
In-hospital Length of Stay | Day 1 (cefiderocol initiation) up to Day 28, death, or discharge (whichever occurs first)
  Length of stay in hospital (days) for participants with infections treated by cefiderocol will be reported.
Length of Stay in Intensive Care Unit (ICU) | Day 1 (cefiderocol initiation) up to Day 28, death, or discharge (whichever occurs first)
  Length of stay in ICU (days) for participants with infections treated by cefiderocol will be reported.
Length of Invasive Ventilation | Day 1 (cefiderocol initiation) up to Day 28, death, or discharge (whichever occurs first)
  Length of invasive ventilation (days) for participants with infections treated by cefiderocol will be reported.
All-cause In-hospital Mortality | Day 14, Day 28
  All-cause in-hospital mortality will be reported after cefiderocol initiation.
Cause of Death | Day 1 (cefiderocol initiation) through Day 28
  The relation of death to the reference infection, as reported in the medical notes, will be reported.
Rate of Microbiological Eradication | Day 1 (24 hours post cefiderocol initiation) through Day 28
  The rate of eradication of carbapenem-resistant GNIs will be reported as the percent microbiological eradication among participants with blood stream infections (BSIs) and complicated urinary tract infections (cUTIs)/UTIs from 24 hours of cefiderocol initiation until Day 28. BSI microbiological eradication will be defined as the absence of a positive follow-up blood culture, in which the same organism as the initial blood culture was obtained. Any positive blood cultures drawn within 24 hours of the initial positive culture will be considered as the same episode. cUTI/UTI microbiological eradication will be defined as an absence of a positive follow-up culture of the same organism as the initial infection obtained.
Severity of Illness | Day 1 (cefiderocol initiation) through Day 28
  The severity of illness at the time of cefiderocol administration at baseline will be described by a Sequential Organ Failure Assessment (SOFA) Score, quickSOFA (qSOFA) score, level of organ support, and presence of septic shock. The SOFA score for participants in ICU or qSOFA score for participants outside ICU will be reported for days -3, 0, and 7 in relation to the date of cefiderocol initiation.
Number of Participants With Adverse Drug Reactions (ADRs) | Up to 28 days post-treatment completion with cefiderocol, death, or discharge (whichever occurs first)
  The number of participants with serious and non-serious adverse events with explicit attribution to cefiderocol (ADR) will be reported.
Number of Participants Experiencing Resolution of Infection or Clinical Cure After Prolonged Treatment With Cefiderocol | Day 1 (cefiderocol initiation), every 10 days up to Day 60

CONTACTS AND LOCATIONS:
Locations (55):
- Spain (55):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital General Universitario de Alicante Doctor Balmis, Alicante
  - Hospital Universitario de Torrevieja, Alicante
  - Hospital Universitario San Juan de Alicante, Alicante
  - Hospital Vega Baja de Orihuela, Alicante
  - Hospital Universitario Torrecardenas, Almeria, Almería
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario de Cruces, Bilbao
  - Hospital Universitario de Burgos, Burgos
  - Hospital General Universitario de Ciudad Real, Ciudad Real
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario de Guadalajara, Guadalajara, Guadalajara
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario de Jerez, Jerez de la Frontera
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria
  - Hospital Central de La Defensa Gómez Ulla, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Fundación Alcorcón, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Infanta Sofía, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Sureste, Arganda del Rey, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Complejo Hospitalario Universitario de Ourense, Ourense
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Quironsalud Palmaplanas, Palma de Mallorca
  - Complejo Hospitalario de Navarre, Pamplona
  - Complejo Hospitalario de Pontevedra, Pontevedra
  - Hospital Universitario de Canarias, La Laguna, Santa Cruz de Tenerife
  - Hospital Universitario Nuestra Señora Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Complejo Hospitalario Universitario de Santiago, Santiago
  - Hospital Público Comarcal de la Merced, Seville
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Virgen de la Salud, Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Universitari de Vic (Consorci Hospitalari de Vic), Vic
  - Hospital Álvaro Cunqueiro, Vigo
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital Univeritario Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Torre-Cisneros J, Almirante B, Martos CF, Rascado P, Lleti MS, Sanchez-Garcia M, Soriano A, Soriano-Cuesta MC, Gonzalez Calvo AJ, Karas A, Sarda J, Verardi S, Ferrer R. Effectiveness and safety of cefiderocol treatment in patients with Gram-negative bacterial infections in Spain in the early access programme: results of the PERSEUS study. Eur J Clin Microbiol Infect Dis. 2025 Jun;44(6):1375-1390. doi: 10.1007/s10096-025-05108-6. Epub 2025 Mar 25. PMID 40131647
- [Derived] Torre-Cisneros J, Ferrer R, Martos CF, Sarda J, Gonzalez Calvo AJ, Verardi S, Karas A, Soriano A. Cefiderocol treatment for patients infected by Stenotrophomonas maltophilia, Burkholderia cepacia complex and Achromobacter spp.: subgroup analysis from the PERSEUS study. Eur J Clin Microbiol Infect Dis. 2025 Jun;44(6):1367-1374. doi: 10.1007/s10096-025-05109-5. Epub 2025 Mar 24. PMID 40126766